CLINICAL TRIAL: NCT05708092
Title: NeuroResource Facilitation for Improved Re-Entry Outcomes for Offenders With Brain Injury: A Multi-Site Randomized Controlled Trial
Brief Title: NRF for Improved Re-Entry Outcomes for Offenders With Brain Injury (Brain Injury RE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Brain Injury Association of Pennsylvania (Unknown)
Responsible Party: Principal Investigator, Maria Kajankova, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-21-00561; 2020-75-CX-0007 (Other Grant/Funding Number: National Institute of Justice)
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Brain Injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only the follow up data collector will be blinded to the randomization assignment of all participants. At the beginning of each interview, the participant will be instructed to not share whether they were assigned to a NRF or SOC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NeuroResource Facilitation (Active Comparator): As part of the NRF intervention group, participants will receive specialized care management, both in prison and after the participant goes home. While in the State Correctional Institution (SCI), participants will meet weekly to monthly depending on resource needs, and how close participant is to release with a NeuroResource Facilitator in person who will help participants to understand more about their challenges. Participants may also be referred to a group run by the Facilitator in conjunction with staff from the prison. The facilitator will also tell the participant about resources that are available to help after the participant's release and help participants get connected to them.
  Interventions: Behavioral: NeuroResource Facilitation (NRF)
- Standard of Care (No Intervention): As part of the SoC, participants will receive the re-entry services normally receive if not in the study including (but not limited to) Treatment Services, Educational and Vocational Training, Mental Health Management, Reentry and Transitional Services, Population Management and Community Corrections.

INTERVENTIONS:
Behavioral: NeuroResource Facilitation (NRF) — NRF is defined as a specialized service that promotes access to services and coordinates care specific to the needs of individuals with brain injury.
  Possible resources include vocational services, medical assistance, Social Security (SSI or SSDI if appropriate), and other organizations that can support reentry. If needed to gain access to services and organizations, the facilitator will also provide participants with a summary that includes results from brain injury screenings questionnaire, neurocognitive (thinking abilities) tests, and symptoms. The researchers will share information and coordinate with prison and parole staff about participation in the study. Participant's information will also be shared with resources that could help participants after release, such as funding sources and brain injury services. After release from SCI, the NRF facilitator will assist the participant with all the preparation and logistics associated with the resources the participant applied to.
  Arms: NeuroResource Facilitation

SUMMARY:
The purpose of this study is to evaluate the effectiveness of NeuroResource Facilitation, a novel/innovative intervention, in reducing recidivism in offenders with brain injury (BI).

DETAILED DESCRIPTION:
The prevalence of brain injury (BI) is significantly greater in justice-involved populations, and a substantial proportion of prisoners have likely experienced a BI during their lifetime. A history of BI has a statistically significant association with increased use of correctional, medical and psychological services including crisis intervention; an increased frequency of institutional misconducts; and higher recidivism rates. Brain injury in justice-involved populations is frequently undiagnosed, and therefore untreated, which contributes to the cycle of recidivism. Identifying BI opens up new resources to ex- offenders that can more effectively help them to become productive in their lives in the community. In partnership with the Icahn School of Medicine at Mount Sinai, the Brain Injury Association of Pennsylvania, and the Pennsylvania Department of Corrections (PADOC), this project will implement a randomized clinical trial to determine if a case management intervention called Neurorehabilitation Facilitation (NRF) is effective in reducing recidivism by ten percent in offenders with acquired BI. Offenders in two Pennsylvania prisons (State Correctional Institution (SCI) sites in PA, SCI Phoenix, SCI Chester, SCI Frackville, and SCI Mahanoy) will be screened for BI and cognitive impairment, and those who screen positive will be randomized to receive the intervention or to receive standard of care (SoC). Two thirds of those randomized will receive the intervention and the remaining one third will serve as controls. All participants will be followed for up to three years following their release to examine the immediate and long-term reduction in recidivism.

The primary hypothesis is that NRF, as compared to SoC, will result in a 10% reduction in average 1-year recidivism, estimated by the 2013

Department of Corrections (DOC) report as 35-38%. Understanding that additional factors will contribute to the effect of NRF, the required sample was based on the primary analysis, a logistic regression of the binary response variable recidivism, adjusted for additional independent variables (described below) in the model with estimated R-squared=0.10. An effect size of 10% reduction corresponds to an odds ratio in this model of 0.643. With two thirds (67%) of cases randomized to NRF, and one third (33%) randomized to SoC, a total sample of N=688 provides 80% power at alpha set at 0.05. Anticipating that there will be a loss of approximately 10% of randomized cases to attrition, N=764 cases will be randomized, with n=509 cases randomized to NRF and 255 randomized to SoC.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Proficient in English
* History of brain injury (OSU-TBI-ID)
* Significant cognitive impairment (RBANS and Trails A&B)
* Within 6 months of release
* Returning to 6 county area (Bucks, Chester, Delaware, Montgomery, Philadelphia and Schuylkill)

Exclusion Criteria:

* Non-English Speaking
* Under 18 years old

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1032 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Recidivism | at year 1
  According to the PADOC, rearrest is measured as the first instance of arrest after inmates are released from state prison and reincarceration is measured as the first instance of returning to state prison after an offender is released from state prison.
  Overall recidivism is measured as the first instance of any type of rearrest or reincarceration after inmates are released from state prison.
Number of Recidivism | at year 3
  According to the PADOC, rearrest is measured as the first instance of arrest after inmates are released from state prison and reincarceration is measured as the first instance of returning to state prison after an offender is released from state prison.
  Overall recidivism is measured as the first instance of any type of rearrest or reincarceration after inmates are released from state prison.

SECONDARY OUTCOMES:
Number of Productive Activities Hours | up to 36 months post release
  Productive Activities Hours include competitive employment (hours worked), and volunteer work (hours worked), brain injury clubhouses (hours attended), vocational training program (hours attended), and education (hours attended).
Number or Participants Engaged in Productive Activity | up to 36 months post release
  The number of participants who engage in vocational training program or education activity at end of program.
Number of Participants Engaged with Services | up to 36 months post release
  Engagement with Services. Engagement with Services includes community-based specialized NeuroRehabilitation services (physical therapy, occupational therapy, speech therapy, cognitive rehabilitation therapy, neuropsychology), and vocational rehabilitation services (job development, job placement, job coaching).
Number of Participants Connected to Health/Medical Resources | up to 36 months post release
  The connection to Health/Medical resources will also be measured, "safety net" resources (SNAP, MA, SSI, food bank, etc).
Number of participants in Community Support | up to 36 months post release
  Community Support - Participation in support groups and recovery resources, including religious activities, recreation, and access to transportation.
Number of Participants in Stable Housing | up to 36 months post release
  Community Support - whether the ex-offender has stable housing
Number of Parole Obligations Met | up to 36 months post release
  Parole Obligations - the extent to which the ex- offender has satisfied the obligations of Parole will be tracked, such as whether they have completed all mandated treatment
Number of Participants Discharged from Supervision | up to 36 months post release
  Number of participants that have been or (are likely to be) discharged from supervision.
Date of Reception | up to 36 months post release
  The day on which an individual was initially received into the custody
Date Committed | up to 36 months post release
  The day on which an individual was committed to sentenced
Date of entry into Department of Corrections | up to 36 months post release
  The day on which an individual was admitted into the Department of Corrections
Number of Participants with particular Classification of Offense | up to 36 months post release
  Number of Participants with particular Classification of Offense as listed by the Department of Corrections
Number of participants who are Guilty but mentally ill | up to 36 months post release
  Number of participants who are guilty but mentally ill
Number of Participants Recommended for aftercare | up to 36 months post release
  Number of Participants Recommended to receive aftercare
Status of Participants after Program completion | up to 36 months post release
  Status of Participants after Program completions as determined by the Department of Corrections
Program category | up to 36 months post release
  Program category as as determined by the Department of Corrections

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kajankova, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Brain Injury Association of Pennsylvania, Carlisle, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals should be directed to maria.kajankova@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link tbd).